CLINICAL TRIAL: NCT05206045
Title: Evolution of the SURvival of Patients With SEzary Syndrome (SS) Over the 1998-2020 Period and Its Association With the Early Use of Therapeutic Monoclonal Antibodies
Acronym: SURPASSe
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211592
Record Dates: First submitted 2022-01-24; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Sezary Syndrome; Cutaneous T Lymphoma
MeSH Terms: conditions — Sezary Syndrome | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Sezary syndrome: Adult patient with Sezary syndrome diagnosed between 1998 and 2020
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Standard of care for patients with Sezary Syndrome

SUMMARY:
Sezary syndrome (SS) is a rare, aggressive and advanced form of cutaneous T lymphoma with a poor prognosis (5-year survival rate varying between 24% and 52%). The treatments are only suspensive with short-term remissions. For the past fifteen years, therapeutic approaches have been based on depleting monoclonal antibodies (anti-CD52, anti-CCR4, anti-KIR3DL2, anti-CD70), or antibody-drug conjugates (anti-CD30). But while the efficacy of mogamulizumab on progression-free survival was reported in the phase III study, no study on a large cohort has compared the current overall survival of patients with Sezary syndrome to that before the era of monoclonal antibodies. In this context, we propose to report a large series of patients with Sézary syndrome in order to compare the current survival of patients with that of the pre-monoclonal antibodies era (1998-2003).

The objective of this study is to assess the evolution of the overall survival of patients with Sezary syndrome since the early use of therapeutic monoclonal antibodies. The underlying hypothesis of this study is that the use of therapeutic monoclonal antibodies has improved the prognosis of these patients. Patients included in this retrospective study are patients with a Sezary syndrome diagnosed between 1998 and 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Patient with Sezary Syndrome diagnosed between 1998 and 2020

Exclusion Criteria:

1. Patient opposition to research
2. Patient under guardianship or curatorship, unable to express opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with Sézary syndrome diagnosed between 1998 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | at 5 years

SECONDARY OUTCOMES:
Overall survival | at 10 years
Overall survival | at 15 years
Sezary syndrome specific survival | at 5 years
Sezary syndrome specific survival | at 10 years
Sezary syndrome specific survival | at 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-Louis, Service de Dermatologie, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bozonnat A, Beylot-Barry M, Dereure O, D'Incan M, Quereux G, Guenova E, Perier-Muzet M, Dalle S, Grange F, Viguier MA, Ram-Wolff C, Feldmeyer L, Beltraminelli H, Bonnet N, Amatore F, Maubec E, Franck N, Machet L, Chasset F, Brunet-Possenti F, Bouaziz JD, Battistella M, Donzel M, Pham-Ledard A, Bejar C, Moins-Teisserenc H, Mourah S, Saiag P, Hainaut E, Michel C, Bens G, Adamski H, Aubin F, Boulinguez S, Joly P, Tedbirt B, Templier I, Troin L, Montaudie H, Ingen-Housz-Oro S, Faiz S, Mortier L, Dobos G, Bagot M, Resche-Rigon M, Montlahuc C, Serret-Larmande A, de Masson A; Cutaneous Lymphomas French Study Group. Real-life efficacy of immunotherapy for Sezary syndrome: a multicenter observational cohort study. EClinicalMedicine. 2024 Jun 21;73:102679. doi: 10.1016/j.eclinm.2024.102679. eCollection 2024 Jul. PMID 39007062